CLINICAL TRIAL: NCT03716401
Title: Prognostic Imaging Biomarkers for Diabetic Kidney Disease
Acronym: iBEAt
Status: Recruiting | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: University of Exeter (Other); University Hospital, Bordeaux (Other); University of Bari (Other); University of Turku (Other); Lund University (Other); Swiss Institute of Bioinformatics (Unknown)
Responsible Party: Principal Investigator, Steven Sourbron, Lecturer, University of Leeds
Other Study IDs: 219542
Record Dates: First submitted 2018-03-01; First posted 2018-10-23 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Kidney Disease
Keywords: Magnetic Resonance Imaging; Ultrasound Imaging; Biomarkers; Prognosis
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Magnetic Resonance Imaging; Ultrasonography; Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and urine samples will be collected from all study participants, including serum, plasma, DNA, and RNA samples. A first morning and additional urine void are requested by all participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Bari: Biopsy Arm: All study participants will undergo a baseline MRI and US and corresponding blood and urine sample collection. This will be followed up annually for additional blood and urine samples.
  Additionally, participants at the Bari site will have an additional renal biopsy at baseline.
  Interventions: Diagnostic Test: MRI (magnetic resonance imaging); Diagnostic Test: US (ultrasound); Procedure: Renal Biopsy
- Bordeaux: MRI Follow-up arm: All study participants will undergo a baseline MRI and US and corresponding blood and urine sample collection. This will be followed up annually for additional blood and urine samples.
  Additionally, participants at the Bordeaux site will have an additional ultrasound US and MRI in Follow-up year 2.
  Interventions: Diagnostic Test: MRI (magnetic resonance imaging); Diagnostic Test: US (ultrasound)
- Exeter: Microvascular arm: All study participants will undergo a baseline MRI and US and corresponding blood and urine sample collection. This will be followed up annually for additional blood and urine samples.
  Participants at the Exeter site will undergo microvascular measurements including estimating glycocalyx thickness at baseline and at 2 years follow-up.
  Interventions: Diagnostic Test: MRI (magnetic resonance imaging); Diagnostic Test: US (ultrasound); Diagnostic Test: Microvascular Assessment
- Leeds: Microstructure MRI arm: All study participants will undergo a baseline MRI and US and corresponding blood and urine sample collection.
  Participants at the Leeds' site will have an extended MRI scan at baseline including novel microstructure MRI measurements.
  Interventions: Diagnostic Test: MRI (magnetic resonance imaging); Diagnostic Test: US (ultrasound)
- Turku: PET arm: All study participants will undergo a baseline MRI and US and corresponding blood and urine sample collection. This will be followed up annually for additional blood and urine samples.
  Additionally, participants at the Turku site will undergo a renal Positron Emission Tomography (PET) scan at the baseline timepoint.
  Interventions: Diagnostic Test: MRI (magnetic resonance imaging); Diagnostic Test: US (ultrasound); Diagnostic Test: Positron Emission Tomography (PET)

INTERVENTIONS:
Diagnostic Test: MRI (magnetic resonance imaging) — An MRI (or magnetic resonance imaging) scan is a radiology technique that uses magnetism, radio waves, and a computer to produce images of body structures. The MRI scanner is a tube surrounded by a circular magnet.
Diagnostic Test: US (ultrasound) — An ultrasound scan is a medical test that uses high-frequency sound waves to capture live images from the inside of the body.
  Other Names: Sonography
Procedure: Renal Biopsy — A kidney biopsy involves taking one or more tiny pieces (samples) of the kidney to look at with special microscopes. The microscopes make it possible to see the samples in greater detail.
  Other Names: Kidney biopsy; percutaneous renal biopsy
  Groups: Bari: Biopsy Arm
Diagnostic Test: Positron Emission Tomography (PET) — Positron emission tomography (PET) uses small amounts of radioactive materials called radiotracers, a special camera and a computer to help evaluate organ and tissue functions. By identifying body changes at the cellular level, PET may detect the early onset of disease before it is evident on other imaging tests.
  Other Names: PET scan
  Groups: Turku: PET arm
Diagnostic Test: Microvascular Assessment — Glycocalyx (a network of membrane proteoglycans and glycoproteins lining all blood vessels) thickness is non-invasively estimated from video clips of sublingual vessels captured using a hand held microscope. Glycocalyx is vital for vascular health; perturbations in the glycocalyx are thought to contribute to numerous vascular health complications including DKD.
  Groups: Exeter: Microvascular arm

SUMMARY:
Diabetic kidney disease (DKD) is a common complication of diabetes, and is now the most common form of chronic kidney disease. DKD is the leading cause of kidney disease requiring dialysis or kidney transplantation, and its global incidence and prevalence have reached epidemic levels. While the risk of developing DKD can be ameliorated by tight blood glucose and blood pressure control, it is not fully preventable and once established DKD cannot be cured. Therefore many patients are left with poor and worsening health and with increased mortality risk. Developing new ways to treat DKD requires healthcare professionals to be able to identify those patients most in need of treatment.

One promising approach for identifying patients that are at risk is the use of imaging measurements (called "biomarkers") derived from Magnetic Resonance Imaging (MRI) and Ultrasound (US) of the kidneys. Evidence from early studies shows that such imaging biomarkers can identify underlying problems in DKD such as blood supply, oxygen supply, kidney scarring and kidney function, in ways that are better than those currently available.

The investigators think that imaging biomarkers will improve the identification of patients who are likely to decline from DKD in the short term. The changes found by imaging may even happen before effects on the blood and urine.

The investigators plan to test this hypothesis by performing a study observing 500 patients with early stage DKD, recruited in 5 sites across Europe. All patients will have detailed assessment at the start of their involvement, including clinical assessment, blood and urine samples, and MRI and US scans. The investigators will look at whether imaging biomarkers are associated with other measures that predict progression in DKD, and follow patients every year for 3 years (4 years total study participation) to see if the imaging biomarkers predict worsening DKD.

DETAILED DESCRIPTION:
STUDY OVERVIEW

Prognostic Imaging Biomarkers for Diabetic Kidney Disease (iBEAt) is a prospective observational multi-centre collaborative cohort study, conducted in 6 European countries. It will have a first phase with a cross-sectional design (for an association study - primary objective) and a second phase with a longitudinal design (for a prognostic objective - secondary objective).

All 5 recruiting centres will follow the same recruitment criteria and take the same data using a standardised methodology, including demographic, clinical and family history, medication history, blood- and urine samples as well as MRI and US. Annual follow-up visits will occur in years 2,3,4, where the same data will be collected except MRI and US (acquired only at baseline). In addition, each of the centres will acquire additional centre-specific data to address ancillary objectives.

All biofluids will be processed on site, stored temporarily and shipped in batches to a central biobank for central analysis and long-term storage (University of Lund, Malmo, Sweden). Hemoglobin, Hematocrit and HbA1c will be measured locally on fresh blood. A proportion of the biofluids will be analysed centrally to address the objectives. The remainder will be stored for future biomarker validation studies to be determined by the study Steering Committee in line with objectives of the Biomarker Enterprise to Attack DKD (BEAt-DKD).

All data generated by the study will be centralised in anonymised form in an archive hosted by the Swiss Institute of Bioinformatics. Data access will be limited to licensed study investigators and ancillary studies approved by the steering committee. MRI images will be analysed centrally in the University of Leeds to extract the imaging biomarkers.

PRE-SCREENING

Study personnel will be trained to initiate screening at several points in the healthcare system where the opportunity exists to identify potential study participants. Potential participants will be identified by study team staff and/or investigators after reviewing the medical records of patients being seen in clinic or in primary care for diagnosis of kidney disease in the management of their diabetes. Some sites may be selecting participants from pre-defined registries of potential patients. If necessary, a partial waiver of informed consent will be sought from the local ethics board to pre-screen these potential participants as possible, or pre-screening will be performed by the clinical care team in collaboration with the study team staff.

Pre-screening includes but is not limited to review of medical records, appointment schedules and laboratory databases with local primary care or specialty physicians as consistent with local ethics review. Specifically, study team staff and/or investigators will be trained to identify participants who satisfy the inclusion criteria. Study team staff and/or investigators will also be trained to review the medical chart for exclusion criteria.

Once pre-screened and identified, potentially eligible patients will be approached by a clinical caregiver to request permission for a study team member to initiate discussion of the iBEAt study.

SCREENING/CONSENTING VISIT

As an introduction to the iBEAt study, a study team member will meet with a potential participant, assess enthusiasm for the study, and complete an eligibility questionnaire with the potential participant. Eligibility questionnaires will be inclusive of all inclusion and exclusion data points with the exception of clinical laboratory values.

When appropriate, informed consent will be obtained. For this purpose the study team member will review and explain necessary information with the potential participant in accordance with the requirements of the respective ethics review and human subject research regulations. The ethics-approved written comprehensive consent documents will be reviewed. Participants will be asked to provide consent to access their local medical record for clinical data for long-term follow-up (maximum 15 years after completion of the study), to store their anonymised data for at least 50 years for future research, and to store their anonymised samples indefinitely for future analyses.

If informed consent is obtained, a study identification number (Study ID) will be assigned and limited demographic data should be collected, including information to contact the participant if the need arises. A random urine sample will be taken at this point and submitted for local Urine Albumin Creatinine Ratio (UACR) analysis. Baseline study visit 1 (V1) can be scheduled, which should occur within 90 days. The screening/consent visit will last 30min - 2hrs depending on site.

The participant should be provided with urine collection materials for the V1 visit first morning void and advised to arrive in a fasted state (fasting for 8 hours prior to appointment), not to smoke for the 4 hours preceding the assessments, and to avoid strenuous, out of the ordinary exercise in the 24hrs before the visit. Medications (hypoglycaemic) may need to be withheld or altered for the study assessment visits to ensure participant well-being (e.g. omitting morning insulin injection to maintain blood glucose levels) and integrity of the study. If modifications are required, they will be discussed and agreed with the participant during the screening visit (to be detailed in the manual of operations).

BASELINE VISIT (Year 1)

A checklist will be administered for key activities and adherence to instructions and medication plan on the 24hrs before the visit. Blood glucose (fingertip) will be checked at the start of the visit and study assessments will not be performed if blood glucose <3.5mmol/l on arrival or if the participant reports a symptomatic hypoglycaemic event on the morning of the visit prior to arrival.

Participants will be asked to provide a urine sample. Afterwards 69,5mL blood will be collected using Standard Operating Procedures (SOPs) and collection materials provided by the central lab in a kit labelled with the study ID.

The samples will be processed locally. UACR measurement and fresh blood analysis will be performed in the local pathology lab. The rest of the samples will stored temporarily at the lab before shipment to the central lab in Malmo, Sweden. If the analysis of the baseline UACR shows a value that is inconsistent with the previous reading at screening, a 3d urine sample will be obtained at a later stage in line with local practice.

After blood and urine collections patients will receive a standardised snack and drink.

A questionnaire will be administered including demographics and medical history, and local lab values for common blood and urine biomarkers. The answers will be pre-populated before the visit with information from medical records where possible, and checked/completed with the participant. The questionnaire will be administered by an investigator and is not patient-facing.

A brief clinical exam will be performed including height, weight, waist and hip circumference, seated and standing blood pressure.

A routine MRI safety checklist will be completed with the participant, as required by local MRI practice. An MRI scan will be performed, which will take about 1 hour and will involve a contrast agent injection. The scan will be performed by a qualified research radiographer.

After MRI participants will undergo a standard renal ultrasound exam.

FOLLOW-UP VISITS (Year 2, 3, 4)

At the annual follow-up visits, all sites will perform a brief clinical exam and administer study questionnaires, collect local lab values, blood, 1st and 2nd void urine. Patient preparation, monitoring and management during the visit will be the same as for Visit 1 to ensure comparable data as in other centres that acquire blood, urine and US at Visit 1. Questionnaires will be inclusive for follow-up data points of those captured at baseline. The study participant should be advised this visit will take 1.5 - 2 hours.

In order to retain patients that are unable to attend the follow-up visits, a system will be set up to follow them up remotely (eg. by phone), and the study team will request access to their clinical records to determine their progression rates.

LONG-TERM FOLLOW-UP (Years 5-19)

Long-term outcome data may continue to be collected on an annual basis from patient's medical records, for a maximum of 15 years after the last study visit.

DATA HANDLING

The key file containing the link between identifiable patient ID and anonymous study ID will be stored securely at the recruiting site. The file will be destroyed 15 years after the last study visit. All other study documentation and data will be labelled by the study ID only.

All research data will initially be recorded on paper sheets that will be stored safely in the anonymised participant file, which will be kept on record as per standard practice. The data will then be entered manually into an electronic data capture system (RedCap) and securely uploaded to a central server hosted by the Swiss Institute of Bio-informatics.

The recorded US and MRI images will be uploaded anonymously onto a central system hosted by the Swiss Institute of Bioinformatics, and reviewed by a qualified radiologist to check for incidental findings. If an incidental finding is recorded the radiologist will act according the standard clinical practices and contact the referring physician, who can then set up a management plan.

The MRI images will be processed by a trained member of the research team at Leeds University to extract the relevant imaging biomarkers. For this purpose the anonymised images will be stored temporarily on a local university PC for processing in dedicated software. All extracted imaging biomarkers will be uploaded to the participant file in the electronic data capture system RedCap hosted by the Swiss Institute of Bioinformatics. After that the local copy of the images on the University PC will be deleted.

Investigators of the recruiting site will retain access to their centrally archived data. Other selected investigators within the BEAt-DKD project, including industry collaborators, can request and obtain access to the data in accordance with the standard grant agreement of IMI projects. The data can also be made available to other researchers in the future, under conditions laid out by the iBEAT steering committee based on a review of the scientific study objectives.

HANDLING OF BLOOD- AND URINE SAMPLES

Urine and blood samples taken at baseline and follow-up visits will be sent to the local lab for processing and temporary storage. A small sample of blood and urine will be forwarded to the clinical lab for UACR reading and fresh-blood analysis, and those data will be recorded in the participants medical records. Other samples will be stored locally at -80deg awaiting regular shipments to the central biobank in Malmo.

The referring physician will review the locally analysed blood and urine readings for incidental findings and take action according to standard clinical practice if abnormal readings are found.

The central biochemical laboratory (Malmö, University of Lund) will prepare kits with sample collection and processing materials for each patient labelled and bar-coded with the study ID, and also arrange shipment from the recruiting site to Malmö. All samples will be stored in Malmö under secure conditions and monitored with a dedicated electronic sample tracking system. A small volume of blood and urine will be analysed in Malmö for known clinical biomarkers according to standardised methods, and the remainder will be stored for future analyses by BEAt-DKD investigators. The samples will also remain available for secondary research provided approval is granted by the iBEAT steering committee.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis Diabetes Type 2;
* eGFR >= 30 ml/min/1.73m2;
* Able to provide informed consent;
* Age between 18 years and 80 years;
* Unchanged antidiabetic and antihypertensive medication for the past 3 months (not including dose changes).

Exclusion Criteria:

* Transplantation (except corneal);
* On permanent dialysis;
* Significant comorbidities with life expectancy of < 1 year;
* Use of investigational drug within 1 month prior to screening;
* Known clinical history of urinary obstruction on renal US: either post-voiding residue over 100 ml, or pyelectasis;
* Known clinical history of aortic endoprosthesis at the renal level;
* Current pregnancy;
* History of Hepatitis B or Hepatitis C +;
* Use of antiretroviral medication;
* Known current or clinical history of renal or urinary tract malignancy;
* Concurrent other renal disease (suspected or proven);
* Cirrhotic liver disease, or non-cirrhotic chronic liver disease where ALT >2 x upper limit of normal;
* Current metastatic malignancy;
* Current malignancy with expected survival < study follow up period (4 years);
* Melanomatous skin cancer < 5 years ago (fully resected melanoma >5 years ago, i.e. surgical cure, can be recruited);
* Any other significant disease or disorder which, in the opinion of the investigators, may either put the patient at risk because of participation in the study, or may influence the result of the study, or the patient's ability to participate in the study;
* Cochlear Implant;
* Aneurysm Clips;
* Neurological stimulator;
* Implanted cardiac devices (ICD, PPM, loop recorders, or any others);
* Metal heart valve;
* History of metal foreign bodies in orbits;
* Other implanted metal device which prevents MR imaging;
* Known allergy to Gadolinium contrast;
* Claustrophobia;
* Weight exceeding 250 kg;
* [Bari arm] Absolute contraindications to percutaneous renal biopsy;
* [Bari arm] Bleeding diathesis;
* [Bari arm] Severe uncontrolled hypertension;
* [Bari arm] End stage renal disease with small hyperechoic kidneys;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is the goal of this study to be as inclusive of Type 2 Diabetes as possible, to create a heterogeneous population of participants in the effort to subcategorize to the greatest extent possible for cross-sectional analysis and potential biomarker identification.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2038-09-01 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional (multi-centre collaboration) | 2 years
  MRI biomarkers will be combined with fluid-based biomarkers to discover radiomics features that correlate with renal function

SECONDARY OUTCOMES:
Longitudinal (multi-centre collaboration) | 4 years
  MRI biomarkers will be combined with patient follow-up data to discover radiomics features that correlate with disease progression

OTHER OUTCOMES:
Turku PET Cohort - Renal Blood Flow | 2 years
  Renal Blood Flow measured by Water-labelled PET/MRI
Bari Biopsy Cohort - Total number of glomeruli | 2 years
  Total number of glomeruli measured on renal histopathology
Leeds Microstructure MRI Cohort - Novel biomarkers of renal microstructure | 2 years
  Novel biomarkers of renal microstructure measured with Diffusion Tensor Imaging and 3D Dynamic Contrast-Enhanced MRI
Bordeaux MRI Follow-up Cohort - two-year rate of change in MRI biomarkers and radiomic signatures | 4 years
  Two-year rate of change in MRI biomarkers and radiomic signatures
Exeter Microvasculature Assessment Cohort - Thickness of the sublingual glycocalyx | 4 years
  Thickness of the sublingual glycocalyx as measured by Glycocheck imaging

CONTACTS AND LOCATIONS:
Overall Officials: Steven sourbron, Study Chair — University of Leeds
Locations (7):
- Turun Yliopisto, Turku, Finland
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France
- Università degli Studi di Bari Aldo Moro, Bari, Apulia, Italy
- Lund University Diabetes Centre, Malmo, Sweden
- Swiss Institute of Bioinformatics, Lausanne, Switzerland
- United Kingdom (2):
  - University of Exeter, Exeter
  - University of Leeds, Leeds

REFERENCES:
- [Background] Grenier N, Merville P, Combe C. Radiologic imaging of the renal parenchyma structure and function. Nat Rev Nephrol. 2016 Jun;12(6):348-59. doi: 10.1038/nrneph.2016.44. Epub 2016 Apr 12. PMID 27067530
- [Derived] Gooding KM, Lienczewski C, Papale M, Koivuviita N, Maziarz M, Dutius Andersson AM, Sharma K, Pontrelli P, Garcia Hernandez A, Bailey J, Tobin K, Saunavaara V, Zetterqvist A, Shelley D, Teh I, Ball C, Puppala S, Ibberson M, Karihaloo A, Metsarinne K, Banks RE, Gilmour PS, Mansfield M, Gilchrist M, de Zeeuw D, Heerspink HJL, Nuutila P, Kretzler M, Welberry Smith M, Gesualdo L, Andress D, Grenier N, Shore AC, Gomez MF, Sourbron S; BEAt-DKD consortium. Prognostic imaging biomarkers for diabetic kidney disease (iBEAt): study protocol. BMC Nephrol. 2020 Jun 29;21(1):242. doi: 10.1186/s12882-020-01901-x. PMID 32600374
- See also: Project website — https://www.beat-dkd.eu/